CLINICAL TRIAL: NCT02333708
Title: Study of Circulating Microparticles in Giant Cell Arteritis
Acronym: MicroGiant
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 2013-A00273-44
Record Dates: First submitted 2015-01-05; First posted 2015-01-07 (Estimated); Last update posted 2022-03-09 (Actual); Status verified 2016-09

CONDITIONS: Giant Cell Arteritis; Acute Phase
MeSH Terms: conditions — Giant Cell Arteritis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (3):
- GCA group
  Interventions: Other: Blood sample
- Inflammatory syndrome (without GCA) group
  Interventions: Other: Blood sample
- Without inflammatory syndrome and without GCA group
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: Blood sample

SUMMARY:
To demonstrate that microparticles (MPs), having a powerful procoagulant potential, are in larger amounts in the blood of patients with histologically proven giant cell arteritis (GCA), compared with patients matched for age, sex and with or without inflammatory syndrome.

ELIGIBILITY:
For GCA group:

Inclusion Criteria:

* Men and women ≥ 18 years of age Patient affiliated to social security regimen
* Informed and having signed the consent form to take part in the study.
* Diagnosis of GCA, meeting at least 3 of the following 5 American College of Rheumatology (ACR) criteria for the diagnosis of GCA, including inflammatory syndrome and having

  * Either temporal artery biopsy showing characteristic GCA abnormality
  * Or inflammatory arteritis on imaging examination

Exclusion Criteria:

* Persons under protection of the court or guardianship
* Inability to understand or to follow study procedures
* Dementia
* cancer diagnosed within the previous 5 years (except for non-melanoma skin cancer or in situ carcinoma of the cervix)non-contributory or inconclusive temporal artery biopsy
* Any conditions that might interfere with MPs level: diabetes, recent endo-arterial gesture, current treatment with corticosteroids.
* Participation in another ongoing clinical trial Current anticoagulant therapy
* Active infectious disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: primary and secondary care hospital
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2015-09; Primary Completion 2023-09-16 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Level of microparticles in the blood of patients with histologically proven giant cell arteritis. | Baseline
  Level of microparticles (MPs) in the blood of patients with histologically proven giant cell arteritis (GCA), compared with patients matched for age, sex and with or without inflammatory syndrome.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire Côte de Nacre, Caen, France